CLINICAL TRIAL: NCT05005767
Title: The Adjunctive Effect of Frankincense Extract Gel on Non-Surgical Treatment of Chronic Periodontitis: Clinical and Microbiological Study.
Brief Title: Effect of Frankincense Extract Gel on Non-Surgical Treatment of Chronic Periodontitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Doaa Ahmed Yousef, lecturer at Periodontology, oral medicine, diagnosis and radiology department, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2D
Record Dates: First submitted 2021-07-31; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Chronic Periodontitis
Keywords: chronic periodontitis.; Frankincense; non surgical treatment
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: twenty patients will be randomly be selected and equally divided into Group I: will receive SRP only, group II: will receive SRP and Frankincense extract the gel. Subgingival application of Frankincense extract gel will be performed following initial SRP )day 1) and at 7, and 14 days.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): ten patients with sites suffering from mild chronic periodontitis sites will be treated with scaling and root planing (SRP) only
  Interventions: Procedure: scaling and root planing
- test group (Active Comparator): Ten patients with sites suffering from mild chronic periodontitis. sites will be treated with scaling and root planing (SRP) and subgingival application of Frankincense extract gel
  Interventions: Procedure: scaling and root planing; Procedure: Frankincense extract gel natural herbal product

INTERVENTIONS:
Procedure: scaling and root planing — will receive scaling and root planing only
Procedure: Frankincense extract gel natural herbal product — will receive Scaling and root planing then. Subgingival application of Frankincense extract gel
  Other Names: Scaling and root planing
  Arms: test group

SUMMARY:
This study will evaluate the effect of the subgingival application of Frankincense extract gel as an adjunct to scaling and root planning (SRP) in chronic periodontitis.

DETAILED DESCRIPTION:
: twenty patients will be randomly selected and equally divided into Group I: will receive SRP only, group II: will receive SRP and Frankincense extract the gel. Subgingival application of Frankincense extract gel will be performed following initial SRP )day 1) and at 7, and 14 days. Clinical measurements included pocket depth (PD), bleeding on probing (BOP), and clinical attachment level (CAL). Real-time PCR was carried out to determine the effect of the treatment on Porphyromonas gingivalis (Pg). Clinical measurements and Plaque samples for PCR were recorded at baseline (before treatment), one, and three months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy patients were selected
* patients who had not received any medications for the previous six months that may interfere with periodontal tissue health or healing.
* Patients should demonstrate their ability to maintain good oral hygiene

Exclusion Criteria:

* Smokers and pregnant patients.
* Medically compromised patients and systemic conditions precluding periodontal surgery.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
probing pocket depth | baseline
  probing pocket depth will be recorded at baseline, at site that will be treated
probing pocket depth | 1 month
  probing pocket depth will be recorded at 1 month at the site to be treated
probing pocket depth | 3 month
  probing pocket depth will be recorded at 3 month at the site to be treated
clinical attachment level | baseline
  clinical attachment level will be recorded at baseline,
clinical attachment level | 1 month
  clinical attachment level will be recorded at , 1 month at the site to be treated
clinical attachment level | 3 month
  clinical attachment level will be recorded at 3 months at the site to be treated
bleeding on probing | baseline
  bleeding on probingwill be recorded at baseline, at the site to be treated
bleeding on probing | 1 month
  bleeding on probingwill be recorded at 1, month at the site to be treated
bleeding on probing | 3 month
  bleeding on probingwill be recorded at 3 months at the site to be treated
PCR for Porphyromonas gingivalis count | baseline
  PCR for Porphyromonas gingivalis count be recorded at baseline, at the site to be treated
PCR for Porphyromonas gingivalis count | 1 month
  PCR for Porphyromonas gingivalis count be recorded at 1, and month at the site to be treated
PCR for Porphyromonas gingivalis count | 3 month
  PCR for Porphyromonas gingivalis count be recorded at 3 months at the site to be treated

CONTACTS AND LOCATIONS:
Locations (1):
- Doaa Ahmed yousef bayoumi, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No